CLINICAL TRIAL: NCT00794755
Title: A Phase III Pilot RCT (Randomized, Controlled Trial) to Assess the Effectiveness of Low Dose Vitamin K1 (200 Micrograms Per Day) on Improving Anticoagulation Control in Unstable Patients on Warfarin
Brief Title: Low Dose Supplementation to Improve Anticoagulation Control With Oral Vitamin K as an Adjuvant to Warfarin Therapy
Acronym: LOCK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Dr. Philip S Wells (Chair, Department of Medicine), Ottawa Hospital Research Institute (OHRI)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OHREB #2008555-01H
Record Dates: First submitted 2008-11-18; First posted 2008-11-20 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-07

CONDITIONS: Coagulation
Keywords: Vitamin K; Vitamin K1 (Phytonadione); Unstable INR; VTE or Thrombosis; Warfarin; Anticoagulation Control; Patients on warfarin with unstable anticoagulation control
MeSH Terms: conditions — Thrombosis | interventions — Vitamin K 1

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin K (Active Comparator)
  Interventions: Dietary Supplement: Vitamin K1 (Phytonadione)
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin K1 (Phytonadione) — Vitamin K1 tablets (100 micrograms per tablet) will be taken by patients randomized to the Vitamin K arm. Dosage is two tablets per day (200 micrograms per day) to be taken with warfarin for the 6 month study period.
  Arms: Vitamin K
Dietary Supplement: Placebo — Lactose-based placebo tablets (identical in appearance to the Vitamin K1 tablets) will be taken by patients randomized to the placebo arm. Dosage is two tablets per day to be taken with warfarin for the 6 month study period.
  Arms: Placebo

SUMMARY:
The main objective of this study is to assess the effectiveness of low dose Vitamin K1 (200 micrograms per day) at improving anticoagulation control in unstable patients on warfarin. This study will also aim to look at effectiveness in the context of genes known to influence warfarin metabolism, variability in the consumption of Vitamin K rich foods, and patient knowledge about warfarin anticoagulation -- factors which have been associated with anticoagulation control and which can influence the effectiveness of this intervention in clinical practice.

DETAILED DESCRIPTION:
A double-blinded placebo controlled pilot RCT assessing the effectiveness of daily supplementation with low dose Vitamin K1 (200 micrograms per day) against placebo at improving anticoagulation control. Previous studies assessing the efficacy of this intervention have been small and further trials are required to evaluate the true effectiveness and safety profile. Furthermore the impact of genetic polymorphisms, known to impact warfarin metabolism, on the effectiveness/safety of this intervention will also be assessed in this study. Demographic and clinical variables as well as potential confounding variables such as variable dietary Vitamin K intake, concomitant interacting medications, and anticoagulation knowledge will be assessed in this study. Given that this is a pilot study we will be looking at recruitment numbers and necessary parameter estimates to determine the number of patients available at our institution for the study. Power analysis will be performed to evaluate the treatment effect size between the placebo and intervention groups.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years old
* Have been on warfarin anticoagulation for at least 9 months
* Have an INR target range of 2.0-3.0
* Have "unstable" anticoagulation control, defined as in the preceding 6 months having at least 3 INRs out of range (>= 3.2 or =<1.8) or at least 3 warfarin dose changes
* Have anticoagulation managed by the Ottawa Hospital Thrombosis Clinic
* Able to provide written, informed consent

Exclusion Criteria:

* Anticipated interruption or termination of warfarin anticoagulation in the next six months for a period of 1 week or greater
* Patient instability in the preceding six months suspected to be due to a) Interruption of warfarin therapy for a period of 1 week or more or b) Significant non-compliance (assessed from patient record)
* Possess a known allergy to Vitamin K or lactose based placebos
* Unable/Refusal to provide written, informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Anticoagulation control -- Point estimates (and standard deviations) for the following variables: Percent time in therapeutic range, standard deviation of INRs, number of INRs outside of therapeutic range, and number of dose changes | At study initiation (for the six month pre-intervention period) and at study completion (after the six-month intervention period)
Recruitment Numbers -- Number of patients deemed eligible, Number of patients solicited, Number of patients screened, Number of patients enrolled, and Number of enrolled patients lost to follow-up | Monthly

SECONDARY OUTCOMES:
Bleeding Events -- Both major and minor as defined by the International Society on Thrombosis and Haemostasis (ISTH) criteria | Over 6 month study period
Recurrent thrombosis | Over six month study period

CONTACTS AND LOCATIONS:
Overall Officials: Philip S Wells, MD, MSc, Principal Investigator — Ottawa Hospital, Ottawa Health Research Institute
Locations (1):
- Ottawa Hospital Thrombosis Clinic, Ottawa, Ontario, Canada